CLINICAL TRIAL: NCT04548193
Title: POW-R Health: Power to Redefine Your Health A Pragmatic Dietary Intervention to Improve Bladder Cancer Survivorship
Brief Title: Behavioral Dietary Intervention for the Improvement of Bladder Cancer Survivorship
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: I 661820; NCI-2020-06639 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 661820 (Other: Roswell Park Cancer Institute); R21CA253910 (NIH)
Record Dates: First submitted 2020-09-09; First posted 2020-09-14 (Actual); Results first posted 2024-08-28 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Stage 0a Bladder Cancer AJCC v8; Stage 0is Bladder Cancer AJCC v8; Stage I Bladder Cancer AJCC v8
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Experimental arm) (Experimental): 6-month Cruciferae intervention
  Interventions: Behavioral: Behavioral Dietary Intervention; Other: Educational Intervention; Other: Questionnaire Administration
- Arm B (Control arm) (Active Comparator): 6-month fruit and vegetable intervention based on NCI guidelines for cancer survivors
  Interventions: Behavioral: Behavioral Dietary Intervention; Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Behavioral: Behavioral Dietary Intervention — Receive live phone call
Behavioral: Behavioral Dietary Intervention — Receive IVR phone messages
Other: Educational Intervention — Receive educational materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial investigates how well a healthy eating program works in improving outcomes in patients with bladder cancer. The behavioral dietary program consists of educational materials, live phone calls, and interactive voice response phone messages. Participating in the healthy eating program may improve eating habits and/or reduce the risk of bladder cancer from coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Develop an evidence-based behavioral intervention to increase cruciferous vegetable intake, with the goal of attaining desirable urinary isothiocyanates (ITC) levels effective for anti-cancer activities.

II. Conduct a feasibility pilot of our dietary behavioral intervention through a hybrid I implementation randomized controlled design in 80 non-muscle invasive bladder cancer (NMIBC) survivors, where the treatment group (n=40) will receive an evidence-based telephone intervention to increase cruciferous vegetable intake and the control group (n=40) will receive a general fruit and vegetable intake intervention based on National Cancer Institute (NCI) guidelines.

SECONDARY OBJECTIVE:

I. To ascertain the level of gene expression changes in urinary exfoliated epithelial cells (due to the intervention) as a surrogate for intermediate efficacy.

EXPLORATORY OBJECTIVE:

I. Engage the clinical care providers of patients enrolled in our intervention to ascertain the barriers and facilitators of intervention implementation within clinical practice through conducting 20 semi-structured interviews.

OUTLINE:

AIM I: Develop an evidence-based behavioral intervention using a systematic process consisting of information gathering, discussion groups, and mock intervention delivery.

AIM II: Patients are randomized to 1 of 2 arms.

ARM A (HEALTHY EATING PROGRAM A): Patients receive mailed educational materials about the importance of consuming cruciferae, setting healthier eating goals, and the importance of keeping track of what they eat. Patients also receive one phone call from study staff to make sure they understood the educational materials received and 11 interactive voice response (IVR) phone messages over 6 months.

ARM B (HEALTHY EATING PROGRAM B): Patients receive mailed educational materials about general fruit and vegetable intake, setting healthier eating goals, and the importance of keeping track of what they eat. Patients also receive one phone call from study staff to make sure they understood the educational materials received and 11 IVR phone messages over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* CANCER PATIENT: Age 18 years old or older (no upper limit)
* CANCER PATIENT: English speaking
* CANCER PATIENT: Diagnosed with stage Tis, Ta, or T1 bladder cancer
* CANCER PATIENT: Resides in the Western New York catchment area
* CANCER PATIENT: Did not receive a partial or radical cystectomy
* CANCER PATIENT: Does not have a prior cancer diagnosis within 12 months of their bladder cancer diagnosis
* CANCER PATIENT: Does not have a subsequent more advanced bladder cancer diagnosis
* CANCER PATIENT: For Roswell Park Cancer Registry only: Bladder cancer diagnosed 2016-2018, 2019-current
* CANCER PATIENT: Participant must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure.
* PHYSICIAN: English speaking
* PHYSICIAN: Physician in a clinic located in the catchment area
* PHYSICIAN: Currently treats bladder cancer patients

Exclusion Criteria:

* CANCER PATIENT: Participants who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* CANCER PATIENT: Participants with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events
* CANCER PATIENT: Adults unable to consent
* CANCER PATIENT: Adults unable to complete study measures in English
* CANCER PATIENT: Individuals who are not yet adults (infants, children, teenagers)
* CANCER PATIENT: Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* CANCER PATIENT: Unwilling or unable to follow protocol requirements
* PHYSICIAN: Unable to complete the study measures in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Yeary, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty nine patients were randomized; 7 participants were subsequently excluded due to death, loss of interest, other medical problems, they underwent a cystectomy, or loss to follow-up. Thus, a total of 42 participants completed both baseline and 6-month follow-up assessments, yielding a retention rate of 86%.
Groups:
- Arm A ( Experimental Arm): 6-month Cruciferae intervention
Period: Overall Study
Arm/Group | Arm A ( Experimental Arm) | Arm B (Control Arm)
Started | 25 | 24
Completed | 22 | 20
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 0 | 1
Not completed — Not eligible. Participant underwent cystectomy in August | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2

BASELINE CHARACTERISTICS:
Population: Baseline analysis was performed on participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Experimental Arm) | Arm B (Control Arm) | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 6 | 14
  >=65 years | 14 | 14 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.8 (9.6) | 68.1 (9.1) | 67.4 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 16 | 14 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 20 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Urinary Isothiocyanates Levels
Description: Will be measured using high performance liquid chromatography (HPLC)-based cyclocondensation assay. The outcome is defined as change from baseline in measured levels. Between-group difference of change from baseline was analyzed using Wilcoxon rank-sum tests.
Time Frame: 6 months
Population: One patient from Arm B (Control arm) missed baseline and another patient from Arm B (Control arm) missed follow up data. Hence, only 18 patients are included in the final analysis
Measure: Mean (Standard Deviation); unit: mM
Groups:
- Arm B (Control Arm): a 6-month fruit and vegetable intervention based on NCI guidelines for cancer survivors
Arm/Group | Arm A (Experimental Arm) | Arm B (Control Arm)
Number analyzed (Participants) | 22 | 18
mM | 10.4 (22.5) | 4.3 (14.1)
Statistical Analysis 1: Comparison: Arm A (Experimental Arm) vs Arm B (Control Arm); Test type: Superiority; p = 0.28, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 6.14, 95% CI 2-sided [-5.72 to 17.99]

2. Primary Outcome: Cruciferae Intake Change
Description: Will be assessed using a questionnaire adapted from Thomson et al. to capture both intake and cooking styles. The outcome is defined as change from baseline in measured levels. Between-group difference of change from baseline was analyzed using Wilcoxon rank-sum tests.
Time Frame: 6 months
Population: One patient missed follow up date and was not included in the final analysis. Hence only 19 patients are included in the arm B(Control arm) for this analysis.
Measure: Mean (Standard Deviation); unit: cups/day
Arm/Group | Arm A (Experimental Arm) | Arm B (Control Arm)
Number analyzed (Participants) | 22 | 19
cups/day | 0.78 (0.87) | 0.058 (1.17)
Statistical Analysis 1: Comparison: Arm A (Experimental Arm) vs Arm B (Control Arm); Test type: Superiority; p = .0054, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.72, 95% CI 2-sided [0.06 to 1.38]

3. Secondary Outcome: Gene Expression
Description: Will be evaluated via ribonucleic acid-sequencing (RNA-seq) as a surrogate for intermediate efficacy, conducted at Roswell Park's Genomics Shared Resource using NextSeq500 platform (Illumina Inc.). Will summarize changes between pre- and post-intervention for both arms and calculate point estimates and their corresponding 95% confidence intervals. Will analyze between-group differences in the change of outcome variables between baseline and post-intervention using ANCOVA.
Time Frame: 6 months
Population: No data was collected for this outcome.
Arm/Group | Arm A (Experimental Arm) | Arm B (Control Arm)
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Cruciferous Vegetable Intake, Cups/Day
Description: Will be evaluated by three non-consecutive 24-hour dietary recalls (two weekdays, one weekday) conducted by trained staff using the interview-administered Nutrition Data System for Research (NDSR). The outcome is defined as change from baseline in measured levels. Between-group difference of change from baseline was analyzed using Wilcoxon rank-sum tests.
Time Frame: 6 months
Population: Cruciferous vegetable intake, cups/day
Measure: Mean (Standard Deviation); unit: cups/day
Arm/Group | Arm A (Experimental Arm) | Arm B (Control Arm)
Number analyzed (Participants) | 22 | 20
cups/day | 1.01 (1.31) | 0.07 (0.92)
Statistical Analysis 1: Comparison: Arm A (Experimental Arm) vs Arm B (Control Arm); Test type: Superiority; p = .0098, Wilcoxon (Mann-Whitney); Mean Difference (Final Values) = 0.94, 95% CI 2-sided [0.24 to 1.65]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse events will be labeled as to whether attributed to behavior intervention or not, classified as mild, moderate, severe, life threatening, or causing death, and reported to Roswell Park IRB and NIH under Institute guidelines.
Arm/Group | Arm A ( Experimental Arm) | Arm B (Control Arm)
All-Cause Mortality (participants affected / at risk) | 0/25 | 1/24
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/24
Other Adverse Events (participants affected / at risk) | 0/25 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-31): https://cdn.clinicaltrials.gov/large-docs/93/NCT04548193/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/93/NCT04548193/ICF_001.pdf